CLINICAL TRIAL: NCT04750304
Title: Evaluation of the Use of an E-health Therapeutic Education Application for Osteoarthritis Patients
Acronym: ARTHe 2
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Openium (Unknown); Caleden (Unknown); Innovatherm (Industry); BPIfrance (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2020 COUDEYRE
Record Dates: First submitted 2021-02-10; First posted 2021-02-11 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-02

CONDITIONS: Osteo Arthritis Knee
Keywords: Osteoarthritis; Gonarthrosis; smarthpone application; e-Health
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Application ARTHe — Patient will use ARTHe Application for 3 months

SUMMARY:
Osteoarthritis is the most common joint disease affecting the joint in a comprehensive and progressive manner. It leads to increasing disability.

The recommendations of recent years favor the non-pharmacological treatment of osteoarthritis including regular physical activity, therapeutic education and weight loss Osteoarthritis population has a low level of physical activity due to a lack of information, motivation and false beliefs related to physical activity and kinesiophobia (fear of movement) A preliminary qualitative study (ARTHe1) evaluating the barriers and levers of the use of an e-health therapeutic education application in patients with osteoarthritis was carried out in order to guide the development of the ARTHe application.

The objective of this study is to have the application tested on a panel of patients in order to assess the benefits of using the application in terms of adherence to the practice of physical activity but also in clinical terms on function and pain, and the satisfaction of the patient

DETAILED DESCRIPTION:
This is a prospective observational study including the evaluation of the use of the ARTH-e application after 3 weeks, 6 weeks and 3 months of use.

Patient recruitment will be done in the PRM department of Clermont-Ferrand University Hospital A subgroup of patients will receive a Garmin VivoSmart 4 connected wristband, which will record intrinsic stress measurement data during the test.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients with osteoarthritis according to the ACR (American College of Rheumatology) criteria, symptomatic and diagnosed before inclusion by a specialist or not.
* Patients with least one knee impairment
* Patients with a smartphone or tablet with at least Android 5 or iOS 11.
* Volunteer patients willing to participate in the study.

Exclusion Criteria:

* Patients with no diagnostic criteria for ACR.
* Patients with comprehension disorders making it impossible to interview and complete questionnaires or use the application.
* Refusal to participate or being already included in a research protocol that could influence the current protocol.
* Patients under guardianship, curatorship or deprived of liberty.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with knee arthritis and using a smartphone
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Excercie adherence | 3 weeks
  Measured with Exercice Adherence Rating Scale (EARS) on 5 point Likert scale, 0= totally agree, 5 = totally disagree
Excercie adherence | 6 weeks
  Measured with Exercice Adherence Rating Scale (EARS) on 5 point Likert scale, 0= totally agree, 5 = totally disagree
Excercie adherence | 3 months
  Measured with Exercice Adherence Rating Scale (EARS) on 5 point Likert scale, 0= totally agree, 5 = totally disagree

SECONDARY OUTCOMES:
Pain with analogic visual scale | 3 weeks, 6 weeks, 3 months
  average pain of the 3 prior days, collected on phone interview with analogic visual scale (0 = no pain, 10 = maximum pain )
Functional evaluation | 3 weeks, 6 weeks, 3 months
  Collected on the phone with Knee injury and Osteoarthritis Outcome Score (KOOS).
  This questionnaire contains 17 statements answering the question "During the last eight days, what was your difficulty with each of the following activities?" ". The responses range from "absent" (0 points) to "extreme" (4 points). The maximum score is 68. A high score is predictive of functional degradation.
Satisfaction questionnaire | 3 months
  Collection after 3 months of use, of the evaluation of the application via a quality questionnaire in 3 parts including the general user experience, closed questions on the user interface and open questions on user expectations, this questionnaire will be sent by email.
Frequency of opening the application per week | From day 1 to 3 months
  Collection of application usage parameters in a codified manner
Frequency of opening the application with on exercice session per week | From day 1 to 3 months
  Collection of application usage parameters in a codified manner
Time spent on the application at each opening | From day 1 to 3 months
  Collection of application usage parameters in a codified manner
Number of sessions carried out on a level before moving to the next level | From day 1 to 3 months
  Collection of application usage parameters in a codified manner
Rating of exercice session (out of 5 stars) | From day 1 to 3 months
  Collection of application usage parameters in a codified manner
Rate of positive responses to questionnaires true / false | From day 1 to 3 months
  Collection of application usage parameters in a codified manner
Average weekly pain level | From day 1 to 3 months
  Average pain level will be asked on the application at most twice a week. Collection of application usage parameters in a codified manner
Daily number of steps | From day 1 to 3 months
  Collection of intrinsic activity data for a subgroup using a connected bracelet Garmin in vivo 4, in a codified manner
Intensity of movement | From day 1 to 3 months
  Intensity of movement per day using Metbolic Equivalebt Task (MET) scale will be collected for a subgroup using a connected bracelet Garmin in vivo 4, in a codified manner
Daily heart rate | From day 1 to 3 months
  Daily average, minimum and maximum heart rate will be collected for a subgroup using a connected bracelet Garmin in vivo 4, in a codified
Daily heart variability | From day 1 to 3 months
  Collection of intrinsic activity data for a subgroup using a connected bracelet Garmin in vivo 4, in a codified manner
Daily energy expenditure in calories | From day 1 to 3 months
  Daily energy expenditure in calories will be collected for a subgroup using a connected bracelet Garmin in vivo 4, in a codified manner

CONTACTS AND LOCATIONS:
Locations (1):
- Clermont-Ferrand University Hospital, Clermont-Ferrand, AURA, France